CLINICAL TRIAL: NCT02662647
Title: Decitabine Based Chemotherapy Followed by Haploidentical Lymphocyte Infusion for Elderly Patients With AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li-Xin Wang, MD. PH.D, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaNGH-H001
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: AML
Keywords: demethylating agent; lymphocyte infusion
MeSH Terms: interventions — Decitabine; Cytarabine; aclacinomycins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCAG plus HLI (Experimental): Patient will be treated with decitabine and modified CAG regimen followed by HLA haploidentical peripheral mononuclear blood cells infusion.
  Interventions: Drug: Decitabine 20 mg/m²/day for 5 days
- DCAG (Experimental): Patient will be treated with decitabine combining modified CAG regimen without other treatments.
  Interventions: Drug: Decitabine 20 mg/m²/day for 5 days

INTERVENTIONS:
Drug: Decitabine 20 mg/m²/day for 5 days
  Other Names: Cytarabine; aclacinomycin

SUMMARY:
Demethylating agent decitabine enhances the immunogenicity of leukemia cells by inducing the expression of cancer testis antigens (CTAs),MHC class I and II molecules,costimulatory molecules and adhesion molecules. The leukemias cells treated by decitabine will become more sensitive to the following adoptive T cell therapy.We proposed a hypothesis that decitabine-based chemotherapy acts in synergestic with haploidentical lymphocyte infusion in eliciting leukemia specific cytotoxic lymphocyte(CTL) and diminishing leukemic cells.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of AML based on 2008 World Health Organization (WHO) classification of myeloid malignancies
* Must have life expectancy >= 3 months
* Must have the ability to observe the efficacy and events
* Must have no accompany therapy(including steroid)
* Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Must have haploidentical donor

DONOR Inclusion Criteria:

* Must have signed the standard informed consent form; if sufficient cryopreserved cells remain from a previous donation, no additional donation or consent is required
* Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Must not have an advanced malignant hepatic tumor
* Must not receive any other forms of chemotherapy after cell infusion during the treatment protocol
* Must not be receiving any other investigational agents within 14 days of first dose of study drug
* Must not have uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Must not be pregnant or breastfeeding; pregnant women are excluded from this study because decitabine is a Category D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine; these potential risks may also apply to other agents used in this study
* Must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine or other agents used in the study
* Must not have a known or suspected hypersensitivity to decitabine
* Must not be human immunodeficiency virus (HIV)-positive and on combination antiretroviral therapy; these patients are ineligible because of the potential for pharmacokinetic interactions with decitabine; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

DONOR Exclusion Criteria:

* Must not have any underlying conditions which would contra-indicate apheresis
* Must not be pregnant

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
complete remission(CR) rate | 3 months

SECONDARY OUTCOMES:
overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang LX, Mei ZY, Zhou JH, Yao YS, Li YH, Xu YH, Li JX, Gao XN, Zhou MH, Jiang MM, Gao L, Ding Y, Lu XC, Shi JL, Luo XF, Wang J, Wang LL, Qu C, Bai XF, Yu L. Low dose decitabine treatment induces CD80 expression in cancer cells and stimulates tumor specific cytotoxic T lymphocyte responses. PLoS One. 2013 May 9;8(5):e62924. doi: 10.1371/journal.pone.0062924. Print 2013. PMID 23671644